CLINICAL TRIAL: NCT01207869
Title: Intratracheal Instillation of Umbilical Cord-derived Mesenchymal Stem Cells as a Rescue Treatment for Severe Bronchopulmonary Dysplasia
Brief Title: Intratracheal Umbilical Cord-derived Mesenchymal Stem Cells for Severe Bronchopulmonary Dysplasia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Bai-Horng Su, MD, PhD., Chairman of Department of Pediatrics, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMR99-104
Record Dates: First submitted 2010-09-11; First posted 2010-09-23 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Bronchopulmonary Dysplasia; Extremely Premature Infants; Severe BPD That Conventional Therapies Has Failed; No Severe Congenital Anomalies; no Severe IVH Neither Cystic PVL
Keywords: Bronchopulmonary dysplasia (BPD); Extremely premature infant; Mesenchymal stem cells (MSCs); umbilical cord
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal stem cells (Experimental): the ucMSCs suspension(3× 106 cells per kg of the patient's weight) will be instilled through a 6 French end-hole catheter inserted into the infant's endotracheal tube
  Interventions: Biological: ucMSCs
- Control (Placebo Comparator): Normal saline
  Interventions: Other: Normal saline

INTERVENTIONS:
Biological: ucMSCs — the ucMSCs suspension(3× 106 cells per kg of the patient's weight) will be instilled through a 6 French end-hole catheter inserted into the infant's endotracheal tube
  Arms: Mesenchymal stem cells
Other: Normal saline — the same amount of ucMSCs suspension will be instilled through a 6 French end-hole catheter inserted into the infant's endotracheal tube
  Arms: Control

SUMMARY:
Mesenchymal stem cells (MSCs) have been reported to be effective to prevent alveolar growth arrest in experimental bronchopulmonary dysplasia (BPD). The aim is to treat the extremely premature infant with severe BPD to establish whether intratracheal instillation of umbilical cord-derived MSCs (ucMSCs) is safe and effective as a rescue treatment for severe BPD.

ELIGIBILITY:
Inclusion Criteria:

* severe BPD, defined by the National Institute of Child Health and Human Development workshop, who conventional therapies (including furosemide and theophylline, and HFO ventilation) has failed

Exclusion Criteria:

* severe congenital anomalies
* severe intraventricular hemorrhage ≥ grade 3 or cystic periventricular leukomalacia.

Ages: 1 Week to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
The relations between the cytokine concentrations in the BAL fluid and PAP. | Up to 20 weeks
  To examine the relations between the cytokine concentrations in the BAL fluid and PAP.

SECONDARY OUTCOMES:
The severity score of BPD ranging from 0 to 6 on the serial chest radiographs | 6 months to 1 year
  The severity score of BPD ranging from 0 to 6 on the serial chest radiographs will be graded by a single radiologist, without knowledge of the infant's identity or clinical course, using the roentgenographic severity scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Bai-Horng Su, MD, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan